# 研究方案

经皮穴位电刺激对全身麻醉下行腹部手术的老年患者术后谵妄及脑电图特征参数的影响:单中心、随机、双盲、平行对照临床试验

研究中心: 西京医院麻醉科

主要研究者: 路志红

~H • O • > \_

方案版本号: V1.0

方案日期: 2023年09月20日

# 方案摘要

| 项目名称 | 经皮穴位电刺激对全身麻醉下行腹部手术的老年患者术后谵妄及 |
|-------------|---------------------------------------|
| | 脑电图特征参数的影响:单中心、随机、双盲、平行对照临床试 |
| | 验 |
| 研究目的 | 探究 TEAS 对全身麻醉下行腹部手术老年患者术后谵妄及其机制 |
| 9176 1113 | 的影响,以验证 TEAS 能否改善腹部手术老年患者 POD 的发生 |
| | 率 |
| TT 索 2几 21. | · · |
| 研究设计 | 单中心、随机、双盲、平行对照临床研究 |
| 病例总数 | 试验组与对照组共 226 例 |
| 病例选择 | 入选标准: |
| | (1) 年龄≥65周岁; |
| | (2) ASA 分级≤ Ⅲ级; |
| | (3) 拟行择期全麻下腹部手术; |
| | , |
| | (4) 手术时长>2h; |
| | (5) 住院时长>3d; |
| | (6) 签署知情同意书。 |
| | TIF AV T- MA |
| | 排除标准: |
| | (1) 有严重中枢神经系统损伤及严重脑血管疾病患者(格拉斯 |
| | 哥-匹兹堡脑功能表现分级(cerebral performance |
| | category, CPC) 评分 3~5 级); |
| | (2) 术前谵妄评定(CAM)阳性; |
| | (3) 无法配合研究者,如精神疾病或语言障碍; |
| | (4) 严重的肝肾功能不全(Child-Pugh 肝功能分级 B、C 级、 |
| | 血肌酐>186 μ mol/L) |
| | (5) 严重的呼吸系统疾病 |
| | (6) 不适宜实施经皮穴位电刺激者,如体内植入电生理装置、 |
| | 穴位部位皮肤感染破损者。 |
| 研究指标 | 1. 主要研究指标:术后 7d 内谵妄发生率(使用 CAM 量表联合 |
| | 3D-CAM 量表) |
| | 2. 次要研究指标: |
| | (1) 术中脑电图 α 波段功率变化; |
| | (2) 术中局部脑氧饱和度最低值和最大降幅; |
| | (3) 术中脑电图爆发性抑制时间; |
| L | 1 \ / - / / / / |

| | (4) 术后住院期间主要并发症发生率(昏迷、卒中、意识状态 |
|------|------------------------------------------|
| | 改变等); |
| | (5) 术后 1d、3d 时阿森斯失眠量表(the AthensInsomnia |
| | Scale ,AIS)和爱普沃斯嗜睡量表(Epworth |
| | SleepinessScale, ESS) 评分; |
| | (6) 术后 1d、3d 时医院焦虑抑郁量表(HADS) 评分; |
| | (7) 术后 1d、3d 时恢复质量问卷调查表(QoR-15) 评分。 |
| 统计方法 | 基线资料描述性统计分析: |
| | 定量资料以均数土标准差或中位数(四分位间距)表示; 定性资 |
| | 料以数量(百分比)表示;定量数据的组间比较使用两独立样本 |
| | t 检验; 重复测量数据采用重复测量方差分析(analysis of |
| | variance, ANOVA); 定性数据的组间比较采用 x 2 检验或 |
| | Fisher 精确概率法;对于不符合正态分布的数据的组间比较,使 |
| | 用 Mann-Whitney U 检验。统计显著性定义为双侧检验 P<0.05。 |
| 研究中心 | 西京医院麻醉科 |
| 研究期限 | 2023.09-2024.07 |

### 一、研究背景

在全球性人口老龄化的背景下,当前我国人口老龄化已成为人口发展的常态,并且人口老龄化的速度明显加快,程度持续加深。随着人口老龄化发展,接受全身麻醉手术治疗的老年患者比例不断增加,老年患者(即 65 岁或以上)是合并术后谵妄(postaction delirium,POD)的高危人群,POD是一种以注意力不集中、思维紊乱和意识水平改变为特征的一过性脑功能障碍综合征<sup>[1,2]</sup>,通常发生于术后数小时至数日内。高龄是 POD 的独立危险因素,根据不同的研究人群和手术类型,POD 发生率为 20%~80%<sup>[3,4]</sup>。POD 不仅会造成住院时间延长,术后并发症增加,甚至会造成永久性的认知功能损害,降低患者的远期生存率和生活质量<sup>[5]</sup>。由于谵妄发生的机制尚不清楚,缺乏有效的治疗策略,因此,预防谵妄的发生发展至关重要。

脑电图(electroencephalogram, EEG)及脑电相关指标是反映大脑意识状态的重要指标,不同麻醉药物及麻醉深度引起不同的 EEG 特征性变化。研究表明<sup>[6-8]</sup>,原始 EEG 与 POD 的发生发展有一定的相关性,并具有潜在的预测 POD 的价值。例如,心脏手术全麻期间较低的前额叶α波段功率与较差的术后认知功能有关,患者年龄越大 EEG 的特征性改变与 POD 的发生越显著 <sup>[9]</sup>。一项在老年人腹部手术中进行的研究也进一步证实了术中 EEG 低α功率与 POD 有关<sup>[10]</sup>。此外,最近的一项研究表明<sup>[11]</sup>,闭眼状态时枕部的α波段相对功率具有中等的辨别能力,与谵妄严重程度和注意力不集中严重程度成反比。

经皮穴位电刺激(transcutaneous electrical acupoint stimulation,TEAS) 疗法是一种新型物理治疗方法,其将电神经疗法与中医针灸穴位相结合,通过穴位将低频脉冲电流输入,在进行穴位刺激的同时施行低频电疗,以达到治疗疾病的目的[12]。中医认为手少阴心经与手厥阴心包经主情志,用于增强睡眠,治疗神经类疾病。神门穴是手少阴心经的穴位之一,有帮助入眠,调节自律神经,补益心气,安定心神等功效;内关穴是手厥阴心包经的常用腧穴之一,可调节神志,治疗神经衰弱、失眠、中风及后遗症。既往研究显示[13],TEAS 刺激双侧内关、神门穴可改善老年髋部手术患者围术期睡眠质量和减少术后谵妄发生率,而对于老年腹部手术患者的研究证据是十分有限的。TEAS 改善 POD 的机制尚未明确,该过程是否伴随着特定脑电生物标志物的变化是未知的,仍需进行更深一步的探索。因此,应特别加强对老年腹部手术患者围术期脑电活动的监测,以期通过对 EEG 的分析给 TEAS 改善 POD 提供一个强有力的证据。

故本研究旨在观察 TEAS 内关、神门穴对围术期老年患者特定脑电生物标志物的影响,从而进一步探究 TEAS 改善 POD 的机制。

二、 研究目的: 探究 TEAS 对全身麻醉下行腹部手术老年患者术后谵妄及其机制的影响,以验证 TEAS 能否改善腹部手术老年患者 POD 的发生率

- 三、 研究设计: 单中心、随机、双盲、平行对照临床试验
- 四、 研究中心: 西京医院麻醉科
- 五、 患者筛选
  - 1. 入选标准:
  - 1) 年龄≥65周岁;
- 2) ASA 分级≤ Ⅲ级;
- 3) 拟行全麻下择期腹部手术;
- 4) 手术时长>2h;
- 5) 住院时长>3d;
- 6) 签署知情同意书。
- 2. 排除标准:
- 1) 有严重中枢神经系统损伤及严重脑血管疾病患者(格拉斯哥-匹兹堡脑功能表现分级(cerebral performance category, CPC)评分 3~5 级);
- 2) 术前谵妄评定(CAM)阳性;
- 3) 无法配合研究者,如精神疾病或语言障碍;
- 4) 严重的肝肾功能不全(Child-Pugh 肝功能分级 B、C 级、血肌酐 $>186 \mu mol/L$ );
- 5) 严重的呼吸系统疾病;
- 6) 不适宜实施经皮穴位电刺激者,如体内植入电生理装置、穴位部位皮肤感染破损者。

#### 六、 研究方案

- 1. 干预措施
- 1) 干预组(EA组): 电针组,在麻醉诱导开始时将电极片贴于内关穴、神门穴处的皮肤上,用经皮穴位电刺激仪(华佗 SDZ-V型,苏州医疗器械厂)持续给予低频疏密波经皮穴位电刺激 30min(电流强度以患者能耐受的最大电流为宜,频率 2/15Hz);
- 2) 对照组(C组): 非电针组,在麻醉诱导开始时将电极片贴于内关穴、神门穴处的皮肤上,不予刺激。
- 2. 穴位定位

1) 内关穴定位:位于前臂掌侧,当曲泽与大陵的连线上,腕横纹上2寸,掌长肌腱与桡侧腕屈肌腱之间:

- 2) 神门穴定位: 腕横纹尺侧端, 尺侧腕屈肌腱的桡侧凹陷处。
- 3. 研究步骤
- 1) 术前准备阶段
- a. 患者进入手术室后再次确认其入选与排除标准,由研究护士打开患者编号对应的信封,确定 患者分组情况:
- b. 连接监护仪常规监测患者的心电图(ECG)、无创动脉血压(NIBP)、脉搏血氧饱和度(SpO2)、呼吸频率(RR);
- c. 开放静脉通路;
- d. 在麻醉诱导开始前接好脑电监测仪,监测 30min 基线脑电活动;
- e. 麻醉诱导开始之前由专人给患者在相应穴位贴上电极贴,连接经皮穴位电刺激仪(华佗 SDZ-V型,苏州医疗器械厂),调整预定参数,测试患者能忍受的最大电流强度,记录患者最佳刺激强度。
- 2) 麻醉诱导阶段
- a. 根据分组不同在诱导时给予相应的干预措施,将麻醉深度指数维持在40-60之间;
- b. 依次注射舒芬太尼 0.3~0.5 μg /kg, 依托咪酯 0.2~0.6mg/kg, 地塞米松 0.1mg/kg, 待患者意识消失 (大声呼唤及用力拍击肩膀无反应, MOAA/S=0), 静脉注射罗库溴铵 0.6-0.9mg/kg, 行气管插管, 气管插管后行机械通气, 采用容量通气模式, 氧流量 1.5L/min, 潮气量为 6~8ml/kg (体重为校正体重), 呼吸频率为 12 次 /min, 气道峰压< 30 mmHg, 呼气末 CO2 分压维持在 35~45 cmH2O。
- 3) 麻醉维持阶段
- a. 维持期瑞芬太尼 4~6ng/ml, 丙泊酚 2~4ug/ml TCI 维持麻醉, 术中根据麻醉深度调整泵注速度;
- b. 术中血压维持在基础值±20%。
- 4) 手术结束阶段
- a. 手术结束时, 停止麻醉药物输注;
- b. 待患者自主呼吸良好,符合拔管指征后拔除气管导管;
- 5) PACU 停留阶段

- a. 拔管后 30min 评估 CAM 量表,若发生谵妄或其它特殊情况详细描述备注;
- b. 当 Aldrete 评分≥9 分时离开 PACU;
- 6) 术后随访观察阶段
- a. 术后 1、3、5、7d 随访评估 CAM 量表及 3D-CAM 量表,查询病例记录术后并发症;
- b. 术后 1d、3d 时随访评估阿森斯失眠量表(AIS 评分)以及爱普沃斯嗜睡量表(Epworth Sleepiness Scale, ESS)评分;
- c. 术后 1d、3d 时随访评估医院焦虑抑郁量表(HADS) 评分;
- d. 术后 1、3d 时随访评估恢复质量问卷调查表(QoR-15) 评分(QoR-15 量表包括身体舒适度、情绪、生理独立性、心理支持、疼痛和术后恶心呕吐等 15 个项目,每项以 0~10 分评分,取总和为最终评估结果);

### 7) 数据采集:

- 1. 脑电图:术前半小时采集静息态 30min 的基线脑电,术中采用脑电收集仪器持续收集麻醉 诱导开始至手术结束的脑电图:
- 2. 脑氧:采用近红外光谱脑氧饱和度监测仪持续监测从麻醉诱导开始至手术结束的脑氧饱和度变化,并记录局部脑氧饱和度最低值和最大降幅。

# 七、 结局指标

- 1. 主要研究指标: 术后 7d 内谵妄发生率
- 2. 次要研究指标:
- (1) 术中脑电图 α 波段功率变化;
- (2) 术中局部脑氧饱和度最低值和最大降幅;
- (3) 术中脑电图爆发性抑制时间(脑电暴发抑制定义为爆发抑制比(burst-suppression ratio,BSR)≥10% ,超过 1 min):
- (4) 术后住院期间主要并发症发生率(昏迷、卒中、意识状态改变等);
- (5) 术后 1d、3d 时阿森斯失眠量表(the AthensInsomnia Scale, AIS)和爱普沃斯嗜睡量表(Epworth SleepinessScale, ESS)评分:
- (6) 术后 1d、3d 时医院焦虑抑郁量表(HADS) 评分;
- (7) 术后 1d、3d 时恢复质量问卷调查表(QoR-15) 评分。

#### 八、 结果分析:

- 1. 术后 7d 内谵妄发生率;
- 2. 脑电图各波段功率谱分析:
- 3. 术中局部脑氧饱和度最低值和最大降幅。

#### 九、 流程图

| 时间点 | 术前<br>1-7d | 麻醉<br>诱导<br>前 | 麻醉<br>诱导<br>开始 | 麻醉诱<br>导开始<br>5~30mi<br>n | 术中 | 手术<br>结束<br>时 | 手术<br>术后<br>30min | 术后<br>1d | 术后<br>3d | 术后<br>5d | 术后<br>7d |
|---|---|---|---|---|---|---|---|---|---|---|---|
| 筛选 | <b>√</b> | | | | | | | | | | |
| 患者基本信息 | <b>√</b> | | | | | | | | | | |
| 知情同意书 | | | | | | | | | | | |
| 血流动力学指标 | | $\sqrt{}$ | $\sqrt{}$ | | $\sqrt{}$ | $\checkmark$ | | | | | |
| 研究干预 | | | | √ | $\sqrt{}$ | | | | | | |
| 脑电监测 | | $\checkmark$ | | √ | $\sqrt{}$ | | | | | | |
| 局部脑氧饱和度<br>监测 | | V | √ | V | <b>V</b> | | | | | | |
| CAM 量表评分 | | | | | | | $\sqrt{}$ | $\checkmark$ | $\sqrt{}$ | | $\checkmark$ |
| 3D-CAM 量表评<br>分 | | | | | | | √ | V | <b>√</b> | V | <b>√</b> |
| 并发症发生率 | | | | | | | | <b>√</b> | <b>√</b> | | |
| AIS 量表评分 | | | | | | | | $\checkmark$ | $\checkmark$ | | |
| ESS 量表评分 | | | | | | | | <b>V</b> | <b>V</b> | | |
| HADS 量表评分 | | | | | | | | | | | |
| QoR-15 量表评分 | | | | | | | | $\checkmark$ | | | |

注: 患者基本信息(姓名、性别、年龄、身高、体重、住院号、BMI)

# 八、样本量

根据既往研究,我们估计 TEAS 组老年患者术后谵妄发生率为 9.6%[19],对照组老年患者术后谵妄发生率为 24.2%,  $\alpha$  =0.05 (双尾),检验效能 1- $\beta$  =0.8 的条件下,计算每组需要 100 名患者,共计 200 例。考虑到 10%脱落率,则最终确定样本量为 226 例,每组 113 例。

# 九、 患者可能的风险与受益

患者可能的风险为麻醉和手术相关的风险。本研究所采用的方案为临床常用麻醉方案,对患者无经济补偿。

#### 十、 随机和盲法

定义 4 或 6 名患者为一个区组,由一名未参与临床麻醉的研究人员采用计算机生成区组随机化结果,分别密封入信封内。待患者入选,由研究护士按相应入选号打开信封,获得分组结果。

本次试验采用双盲设计,对患者、麻醉医生设盲。

#### 十一、安全性

#### 1. 不良事件

研究者将如实记录不良事件的发生,并且判断是否与试验有关,所有不良事件必须追踪至妥善解决。

#### 2. 可能出现的不良事件以及处理办法

本研究可能发生的不良事件包括手术和麻醉相关的不良事件。严重的不良事件定义为导致如下后果之一:死亡,致残,神经损伤。在临床试验期间发生任何严重不良事件,将在24小时内报告研究者及伦理委员会。

#### 十二、病例脱落

#### 1. 脱落的定义

所有填写了知情同意书并筛选合格进入试验的患者,均有权利随时退出临床试验,无论何时何因退出,凡没有完成方案所规定观察周期的受试者,称为脱落病例。

#### 2. 脱落原因

对于任何脱落病例,研究者必须在 CRF 表中填写脱落的原因,一般情况下有 6 种,即不良事件、缺乏疗效、违背试验方案(包括依从性差)、失访(包括受试者自行退出)、被申办者中止和其他。

#### 十三、 数据收集与管理

所有数据均记录于纸质 CRF 中,采集数据储存在相应设备中,所有文件保存于西京医院麻醉科。

#### 十四、 统计学方法

基线资料描述性统计分析:

定量资料以均数±标准差或中位数(四分位间距)表示。定性资料以数量(百分比)表示; 定量数据的组间比较使用两独立样本 t 检验;

重复测量数据采用重复测量方差分析(analysis of variance, ANOVA);

定性数据的组间比较采用 × 2 检验或 Fisher 精确概率法;

对于不符合正态分布的数据的组间比较,使用 Mann-Whitney U 检验。

统计显著性定义为双侧检验 P<0.05。

# 十五、 研究中心

| 中心 | 主要研究者 | 职称 |
|---------|-------|-----------|
| 西京医院麻醉科 | 路志红 | 副主任医师,副教授 |

#### 十六、 研究日期

研究预计于 2023年 09月至 2024年 7月完成。

# 参考文献

[1] Li T, Li J, Yuan L, et al. Effect of Regional vs General Anesthesia on Incidence of Postoperative Delirium in Older Patients Undergoing Hip Fracture Surgery: The RAGA Randomized Trial[J]. JAMA, 2022,327(1):50-58.

- [2] Wildes T S, Mickle A M, Ben A A, et al. Effect of Electroencephalography-Guided Anesthetic Administration on Postoperative Delirium Among Older Adults Undergoing Major Surgery: The ENGAGES Randomized Clinical Trial[J]. JAMA, 2019,321(5):473-483.
- [3] Mei B, Xu G, Han W, et al. The Benefit of Dexmedetomidine on Postoperative Cognitive Function Is Unrelated to the Modulation on Peripheral Inflammation: A Single-center, Prospective, Randomized Study[J]. Clin J Pain, 2020,36(2):88-95.
- [4] Kotekar N, Shenkar A, Nagaraj R. Postoperative cognitive dysfunction current preventive strategies[J]. Clin Interv Aging, 2018,13:2267-2273.
- [5] Jin Z, Hu J, Ma D. Postoperative delirium: perioperative assessment, risk reduction, and management[J]. Br J Anaesth, 2020,125(4):492-504.
- [6] White M F, Tanabe S, Casey C, et al. Relationships between preoperative cortical thickness, postoperative electroencephalogram slowing, and postoperative delirium[J]. Br J Anaesth, 2021,127(2):236-244.
- [7] Giattino C M, Gardner J E, Sbahi F M, et al. Intraoperative Frontal Alpha-Band Power Correlates with Preoperative Neurocognitive Function in Older Adults[J]. Front Syst Neurosci, 2017,11:24.
- [8] Hesse S, Kreuzer M, Hight D, et al. Association of electroencephalogram trajectories during emergence from anaesthesia with delirium in the postanaesthesia care unit: an early sign of postoperative complications[J]. Br J Anaesth, 2019,122(5):622-634.
- [9] Khalifa C, Lenoir C, Robert A, et al. Intra-operative electroencephalogram frontal alpha-band spectral analysis and postoperative delirium in cardiac surgery: A prospective cohort study[J]. Eur J Anaesthesiol, 2023,40(10):777-787.
- [10] Gutierrez R, Egana J I, Saez I, et al. Intraoperative Low Alpha Power in the Electroencephalogram Is Associated With Postoperative Subsyndromal Delirium[J]. Front Syst Neurosci, 2019,13:56.
- [11] Guay C S, Kafashan M, Huels E R, et al. Postoperative Delirium Severity and Recovery Correlate With Electroencephalogram Spectral Features[J]. Anesth Analg, 2023,136(1):140-151.
- [12] Feng B, Zhang Y, Luo L Y, et al. Transcutaneous electrical acupoint stimulation for post-traumatic stress disorder: Assessor-blinded, randomized controlled study[J]. Psychiatry Clin Neurosci, 2019,73(4):179-186.
- [13] 黄俊. 经皮穴位电刺激神门、内关穴对老年髋关节置换术患者睡眠质量及术后谵妄的影响[D]. 湖南师范大学, 2020.

# 附 录

表1 格拉斯哥-匹兹堡脑功能评分

| +‡+ | | | | |
|-----|------|---------|------------------------------------------|----|
| | 等级 | 功能 | 症状。 | 42 |
| | I级 | 脑功能完好 | 患者清醒警觉,有工作和正常生活能力。 | φ |
| | II 级 | 中度脑功能残障 | 患者清醒,可在特定环境中部分时间工作或独立完成日常活动。 | |
| | Ⅲ级 | 严重脑功能残障 | 患者清醒,因脑功能损害依赖他人的日常帮助,至少存在有限的认知力。 | |
| | N级 | 昏迷及植物状态 | 无知觉,对环境无意识,无认知力,不存在与周边<br>环境的语言或心理的相互作用。 | |
| | V级 | 死亡 | 确认的脑死亡或传统标准认定的死亡。 | |

### 附表 2: CAM 评分细则:

# 特征 1: 急性起病

a. 与基础状态相比,患者是否存在精神状态急性改变? 是=1: 不是=2: 不确定=8

b. 如果"是", 请描述变化情况及信息来源

#### 特征 2: 注意力障碍

a. 患者是否存在注意力难以集中?

如注意力容易转移、无法保持连续性随访期间从未发生=1

随访期间偶尔有,轻度=2

随访期间有,很明显=3

不确定=8b

- b. 如果存在注意力不集中,在随访期间是否出现病情减轻或加重等波动? 是=1;不是=2;不确定=8;不适用=9
- c. 如果"是",请描述

# 特征 3: 思维紊乱

a. 患者是否存在思维无序或无连贯性?

如散漫或不相关谈话、不清晰或没有逻辑性的想法或者不可理解的话题转化随访期间从未发生=1

随访期间偶尔有,轻度=2

随访期间有,很明显=3

不确定=8

b.如果存在思维紊乱,在随访期间是否出现病情减轻或加重等波动?

是=1; 不是=2; 不确定=8; 不适用=9

c.如果"是",请描述

# 特征 4: 意识水平改变

a.你如何对患者的整体意识水平进行分级?

正常=1(如患者意识正常,直接进入第5个问题)

警惕性(如高警觉性、对环境刺激敏感、容易不安)=2

嗜睡(嗜睡但可唤醒)=3

昏睡(难以唤醒)=4

昏迷(无法唤醒)=5

不确定=8

b.如果存在意识水平改变,在随访期间是否出现病情减轻或加重等波动?

是=1; 不是=2; 不确定=8; 不适用=9

c.如果"是",请描述

# 特征 5: 定向力障碍

a. 随访期间患者是否出现定向力障碍?

如地点和时间定向障碍随访期间从未发生=1

随访期间偶尔有,轻度=2

随访期间有,很明显=3

不确定=8

b.如果存在定向力障碍,在随访期间是否出现病情减轻或加重等波动?

是=1; 不是=2; 不确定=8; 不适用=9

| c.如果"是",请描述 |
|-------------|
|-------------|

# 特征 6: 记忆力损害

a.随访期间患者是否出现记忆力损害?

如无法记住医院内发生的事件或难以记住说明随访期间从未发生=1

随访期间偶尔有,轻度=2

随访期间有,很明显=3

不确定=8

b.如果存在记忆力损害,在随访期间是否出现病情减轻或加重等波动?

是=1; 不是=2; 不确定=8; 不适用-9

c.如果"是",请描述

# 特征 7: 记忆力损害: 感知障碍

a.随访期间患者是否出现感知障碍?

如幻视、幻听、幻想随访期间从未发生=1

随访期间偶尔有,轻度=2

随访期间有,很明显=3

不确定=8

b.如果存在感知障碍,在随访期间是否出现病情减轻或加重等波动?

是=1; 不是=2; 不确定=8; 不适用=9

c.如果"是",请描述

# 特征 8: 精神躁动

a.随访期间患者是否出现精神活动增加?

如不安、戳床单、频繁换动体位随访期间从未发生=1

随访期间偶尔有,轻度=2

随访期间有,很明显=3

不确定=8

b.如果存在精神躁动,在随访期间是否出现病情减轻或加重等波动?

是=1; 不是=2; 不确定=8; 不适用=9

c.如果"是",请描述

# 特征9: 睡眠-觉醒周期改变

a.与基础状态相比,患者是否存在睡眠觉醒周期改变?

如白天嗜睡、夜间失眠是=1; 不是=2; 不确定=8

b.如果"是",请描述

#### 诊断标准:

- (1)急性起病 1a 或 2b 或 3b 或 4b=1,此标准成立
- (2)注意力 2a=2 或 3, 此标准成立
- (3)思维紊乱 3a=2 或 3, 此标准成立
- (4) 意识水平改变 4a=2、3、4 或 5, 此标准成立

谵妄诊断成立:

满足以下标准(1)+(2)+(3)或(1)+(2)+(4)

# 附表 3:3D-CAM 评分细则:

| 认知功能(引导语:"我要问你一些关于思考和记忆的问题") | 正确 | 错误 | 拒绝 | 无回答 |
|--------------------------------------------|------|----|----|-----|
| 1.请问今年是哪一年? | 1 | 2 | 7 | 8 |
| 2.请问今天是星期几? | 1 | 2 | 7 | 8 |
| 3.请问这里是什么地方?(回答"医院"即为正确) | 1 | 2 | 7 | 8 |
| 以上 1~3 任一问题答案不是"正确"为特征 | 3 阳性 | | | |
| 4.我要读一些数字,请你按照我读的相反的顺序重复一遍,如我 | 1 | 2 | 7 | 8 |
| 说"6-4",你说"4-6",清楚了吗? 第 1 组数"7-5-1" (1-5-7) | | | | |
| 5.第 2 组数是"8-2-4-3" (3-4-2-8) | 1 | 2 | 7 | 8 |
| 6.请从冬季开始,倒着说出季节。最多可以提示 1 次,如冬季 | 1 | 2 | 7 | 8 |
| 之前是哪个季节?逐一记录回答,任意一个季节错误则整个项 | | | | |
| 目错误 | | | | |
| 冬季 | 1 | 2 | 7 | 8 |
| 秋季 | 1 | 2 | 7 | 8 |
| 夏季 | 1 | 2 | 7 | 8 |
| 春季 | 1 | 2 | 7 | 8 |
| 7.从 20 开始,每次减去 3,请连续计算,直到我说停止为 | 1 | 2 | 7 | 8 |
| 止。当受试者停止 X, 提示"X-3 等于多少?"只能提示 1 次 | | | | |
| 20-3 | 1 | 2 | 7 | 8 |
| 17-3 | 1 | 2 | 7 | 8 |
| 14-3 | 1 | 2 | 7 | 8 |

| 11-3 | 1 | 2 | 7 | 8 |
|------------------------------------|------------|----------|----|-----|
| 8-3 | 1 | 2 | 7 | 8 |
| 以上 4~7 任一问题答案不是"正确"为特征 | 正 2 阳性 | ŧ | | |
| 患者主诉的症状 (如果患者回答"是"请询问细节并记录 否 | 是 | 拒绝 | 无意 | 不知道 |
| 答案。如果受试者回答没有任何意义,编码为8) | | | 义 | |
| 8.最近这一天你有没有感到混乱? 1 | 2 | 7 | 8 | 9 |
| 9.最近这一天你有没有感觉到你不在医院? 1 | 2 | 7 | 8 | 9 |
| 10.最近这一天你有没有看到实际不存在的东西? 1 | 2 | 7 | 8 | 9 |
| 以上 8~10 任一问题答案不是"否"为特征 | <br>E 1 阳性 | <u> </u> | | |
| 观察者评估(询问患者上面 1~10 的问题后完成) | | | 是 | 否 |
| 11A.在评估过程中,患者是否出现困倦?(患者实际入睡,但是 | 1 | 2 | | |
| (特征 4) | | | | |
| 11B.在评估过程中,患者是否昏睡或昏迷?(难以唤醒)(特征 4) | 1 | 2 | | |
| 12.患者是否表现为对环境中常规事物过度的敏感亢奋(警觉性 | 增高)?( | (特征 | 1 | 2 |
| 4) | | | | |
| 13.患者是否思维不清晰或不合逻辑,例如讲述与谈话内容无关 | 长的事情 | f(跑 | 1 | 2 |
| 题)?(特征 3) | | | | |
| 14.患者是否谈话漫无边际,例如他/她有无不合时宜的嘤嗦以及 | 及回答ろ | 下切 | 1 | 2 |
| 题? (特征 3) | | | | |
| 15.患者语言是否比平常明显减少?(例如:只回答是/否)(特征 3) | | | 1 | 2 |
| 16.在评估过程中,患者是否不能跟上正常谈论的话题? (特征 2 | 2) | | 1 | 2 |

| 17.患者是否因为环境刺激出现不适当的走神? (特征 2) | | 1 | 2 |
|----------------------------------------|----------|----------------|----|
| 11.芯有足百四为外境制做山塊小坦当的足徑! (付価 2) | | 1 | 2 |
| 18.在评估过程中,患者是否有意识水平的波动?例如开始时作出适当尽 | 反应, | 1 | 2 |
| 然后迷糊地 | | | |
| 睡去(特征 1) | | | |
| 一座云(行征工) | | | |
| 19.在评估过程中,患者是否有注意力水平的波动?例如患者对谈话的专 | 注度 | 1 | 2 |
| 或注意力测试的表现变化很明显?(特征 1) | | | |
| 20.在评估过程中,患者是否有语言表达/思维的变化?例如患者语速时快 | 时 | 1 | 2 |
| 慢?(特征 1) | | | |
| 可收过度 每些红色现在中间 一国民社会工程会工程会工程会工程 | <b>不</b> | Ħ | ᇤ |
| 可选问题:仅特征1没有出现,同时特征2及特征3或特征4出现时 | 否 | 是 | 跳过 |
| 完成 | | | |
| 21.询问对患者情况非常了解的家人、朋友或医护人员:"是否有迹象 | 1 | 2 | 9 |
| 表明:与患者的平时情况相比,患者存在急性精神状态的变化(记忆或 | | | |
| 思维) ?" (特征 1) | | | |
| 22.如果可获得本次住院或以前的 3D-CAM 评估结果,请与之比较, | 1 | 2 | 9 |
| 根据本次新出现的"阳性"条目,确定患者是否存在急性变化(特征 1) | | | |
| 总结:检查在上列中是否出现了 CAM 相应特征 | | | |
| 谵妄诊断条件:特征 1+特征 2+特征 3 或特征 4。 请在判断结果后打: | 谵妄 ‡ | <b></b><br>上谵妄 | |

方案号: XJH-A-20230920

版本号: V1.0 版本日期: 2023-09-20

# 附表 4: Aldrete 评分细则:

| | 自主或遵嘱活动四肢和抬头 | 2 |
|------|-------------------------|---|
| 活动 | 自主或遵嘱活动二肢和有限制的抬头 | 1 |
| | 不能活动肢体或抬头 | 0 |
| | 能深呼吸和有效咳嗽,呼吸频率和幅度正常 | 2 |
| 呼吸 | 呼吸困难或受限,但有浅而慢的自主呼吸,可能用口 | 1 |
| | 咽通气道 | |
| | 呼吸暂停或呼吸微弱,需呼吸器治疗或辅助呼吸 | 0 |
| | 麻醉前±20%以内 | 2 |
| 血压 | 麻醉前±20%~49% | 1 |
| | 麻醉前±50%以上 | 0 |
| | 完全清醒 (准确回答) | 2 |
| 意识 | 可唤醒,嗜睡 | 1 |
| | 无反应 | 0 |
| | 呼吸空气 Spo2≥92% | 2 |
| SpO2 | 呼吸氧气 Spo2≥92% | 1 |
| | 呼吸氧气 Spo2<92% | 0 |

# 附表 6: 雅典失眠量表 (AIS 量表)

| 自测题目 | 0分 | 1分 | 2分 | 3分 | 得分 |
|------------------|---------------|---------|--------|-----------|-----|
| 1、入睡时间(关灯后到睡着的时 | 没问题 | 轻微延迟 | 显著延迟 | 延迟严重或没有睡觉 | |
| 间) | | | | | |
| 2、夜间苏醒 | 没问题 | 轻微影响 | 显著影响 | 严重影响或没有睡觉 | |
| 3、比期望的时间早醒 | 没问题 | 轻微提早 | 显著提早 | 严重提早或没有睡觉 | |
| 4、总睡眠时间 | 足够 | 轻微不足 | 显著不足 | 严重不足或没有睡觉 | |
| 5、总睡眠质量(无论睡多长) | 满意 | 轻微不满 | 显著不满 | 严重不满或没有睡觉 | |
| 6、白天情绪 | 正常 | 轻微低落 | 显著低落 | 严重低落 | |
| 7、白天身体功能(体力活精神) | 足够 | 轻微影响 | 显著影响 | 严重影响 | |
| 8、白天思睡 | 无思睡 | 轻微思睡 | 显著思睡 | 严重思睡 | |
| 注:总分小于4分:无睡眠障碍;总 | <br>总分在 4-6 ⁄ | ): 可疑睡眼 | 民;总分6分 | 以上:失眠。 | 总分: |